CLINICAL TRIAL: NCT02714400
Title: The Impact of Venlafaxine on Apnea Hypopnea Index in Patients With Obstructive Sleep Apnea
Brief Title: The Impact of Venlafaxine on Apnea Hypopnea Index in Obstructive Sleep Apnea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Robert L. Owens, Assistant Professor, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: UCSD141272ARM5-1
Record Dates: First submitted 2016-02-26; First posted 2016-03-21 (Estimated); Results first posted 2020-04-17 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; Arousal threshold; Venlafaxine
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Venlafaxine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Venlafaxine (Active Comparator): 50mg of Venlafaxine before sleep
  Interventions: Drug: Venlafaxine
- Placebo (Placebo Comparator): One piece of placebo before sleep
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Venlafaxine — Venlafaxine 50mg before sleep
  Arms: Venlafaxine
Drug: Placebo — One piece of placebo before sleep
  Arms: Placebo

SUMMARY:
The investigators hypothesis is that obstructive sleep apnea (OSA) patients with a low arousal threshold may wake up too early during a respiratory event, before upper airway muscles can be activated to achieve stable ventilation. Thus, strategies to manipulate the respiratory arousal threshold could potentially improve the quality of sleep and sleep disordered breathing. Agents that raise arousal threshold are therefore likely to benefit some patients with OSA. The overall goal of this project is to determine the importance of the arousal threshold in OSA, determine which patients might benefit from a raised arousal threshold, and test this hypothesis by using pharmacological manipulation of the arousal threshold to achieve this goal.

DETAILED DESCRIPTION:
This study is a randomized double-blinded crossover pilot study. The investigators will test whether Venlafaxine has important effects on the apnea hypopnea index. Venlafaxine is a serotonin-norepinephrine reuptake inhibitor (SNRI) for the treatment of depression and anxiety. Venlafaxine increases serum serotonin level, which may affect arousal threshold. Furthermore, higher serotonin level theoretically may improve muscle tone, including upper airway muscle. Therefore, the investigators hypothesize that venlafaxine may decrease arousal threshold and improve muscle tone, leading to improvement of OSA.

Eligible participants will undergo overnight polysomonography as described below and will receive either Venlafaxine(50 mg 2 hour prior to sleep) or placebo (in random order) followed roughly 7 days later with placebo or donepezil. This aim will allow us to test the impact of Venlafaxine on the apnea hypopnea index.

The change in apnea hypopnea index will be compared in the Venlafaxine groups with the placebo group.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-70 years
* sleep study (with apnea hypopnea index>5)
* Diagnosis of obstructive sleep apnea

Exclusion Criteria:

* Any known cardiac (apart from treated hypertension), pulmonary (including uncontrolled asthma), renal, neurologic (including epilepsy), neuromuscular, or hepatic disease.
* Susceptible to stomach ulcers.
* co-administration of MAO inhibitors intended to treat psychiatric disorders (concurrently or within 14 days of discontinuing the MAO inhibitor); initiation of MAO inhibitor intended to treat psychiatric disorders within 7 days of discontinuing venlafaxine; initiation in patients receiving linezolid or intravenous methylene blue
* Pregnant women.
* History of hypersensitivity to Afrin, Lidocaine (all Aims) or venlafaxine
* History of bleeding diathesis and/or gastrointestinal bleeding.
* Glaucoma and Urinary Retention
* Use of any medications that may affect sleep or breathing.
* Use of any medications that have known interaction with venlafaxine and the interaction may significantly increase the risk of the subject or decrease the therapeutic effect of the medication.
* A psychiatric disorder, other than mild depression; e.g. schizophrenia, bipolar disorder, major depression, panic or anxiety disorders.
* Substantial cigarette (>5/day), alcohol (>3oz/day) or use of illicit drugs.
* More than 10 cups of beverages with caffeine (coffee, tea, soda/pop) per day.
* Desaturations to below 70% lasting greater than 10 seconds in duration per event

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego, San Diego, California, United States

REFERENCES:
- [Background] Eckert DJ, White DP, Jordan AS, Malhotra A, Wellman A. Defining phenotypic causes of obstructive sleep apnea. Identification of novel therapeutic targets. Am J Respir Crit Care Med. 2013 Oct 15;188(8):996-1004. doi: 10.1164/rccm.201303-0448OC. PMID 23721582
- [Background] Carter SG, Berger MS, Carberry JC, Bilston LE, Butler JE, Tong BK, Martins RT, Fisher LP, McKenzie DK, Grunstein RR, Eckert DJ. Zopiclone Increases the Arousal Threshold without Impairing Genioglossus Activity in Obstructive Sleep Apnea. Sleep. 2016 Apr 1;39(4):757-66. doi: 10.5665/sleep.5622. PMID 26715227
- [Background] Deacon NL, Jen R, Li Y, Malhotra A. Treatment of Obstructive Sleep Apnea. Prospects for Personalized Combined Modality Therapy. Ann Am Thorac Soc. 2016 Jan;13(1):101-8. doi: 10.1513/AnnalsATS.201508-537FR. PMID 26569377
- [Background] Edwards BA, Eckert DJ, McSharry DG, Sands SA, Desai A, Kehlmann G, Bakker JP, Genta PR, Owens RL, White DP, Wellman A, Malhotra A. Clinical predictors of the respiratory arousal threshold in patients with obstructive sleep apnea. Am J Respir Crit Care Med. 2014 Dec 1;190(11):1293-300. doi: 10.1164/rccm.201404-0718OC. PMID 25321848
- [Background] Eckert DJ, Younes MK. Arousal from sleep: implications for obstructive sleep apnea pathogenesis and treatment. J Appl Physiol (1985). 2014 Feb 1;116(3):302-13. doi: 10.1152/japplphysiol.00649.2013. Epub 2013 Aug 29. PMID 23990246
- [Derived] Schmickl CN, Li Y, Orr JE, Jen R, Sands SA, Edwards BA, DeYoung P, Owens RL, Malhotra A. Effect of Venlafaxine on Apnea-Hypopnea Index in Patients With Sleep Apnea: A Randomized, Double-Blind Crossover Study. Chest. 2020 Aug;158(2):765-775. doi: 10.1016/j.chest.2020.02.074. Epub 2020 Apr 9. PMID 32278781

RESULTS

PARTICIPANT FLOW:
Groups:
- Venlafaxine First, Placebo Second: 50mg of Venlafaxine before sleep first night
  1 Pill of Placebo before sleep second night
- Placebo First, Venlafaxine Second: 1 Pill of Placebo before sleep first night 50mg of Venlafaxine before sleep second night
Period: First Intervention (1 Day)
Arm/Group | Venlafaxine First, Placebo Second | Placebo First, Venlafaxine Second
Started | 12 | 8
Completed | 12 | 8
Not Completed | 0 | 0
Period: Washout (>4 Days)
Arm/Group | Venlafaxine First, Placebo Second | Placebo First, Venlafaxine Second
Started | 12 | 8
Completed | 12 | 8
Not Completed | 0 | 0
Period: Second Intervention (1 Day)
Arm/Group | Venlafaxine First, Placebo Second | Placebo First, Venlafaxine Second
Started | 12 | 8
Completed | 12 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Age 35-64 years
Groups:
- All Analyzed Participants: All participants who were randomized, completed both study nights, and were included in the analysis.
Arm/Group | All Analyzed Participants
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.8 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 14
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: The Apnea Hypopnea Index
Description: The Apnea hypopnea index is an index used to indicate the severity of sleep apnea. It is represented by the number of apnea and hypopnea events per hour of sleep. The change from baseline in apnea hypopnea index after a single dose of Venlafaxine will be evaluated using overnight polysomnography. An apnea hypopnea index less than five events per hour is considered within normal limits.
Time Frame: Baseline and 7-day follow up
Measure: Mean (Standard Deviation); unit: Events per Hour of Sleep
Arm/Group | Venlafaxine | Placebo
Number analyzed (Participants) | 20 | 20
Events per Hour of Sleep | 40.5 (16.5) | 46.1 (21.9)

2. Primary Outcome: Nadir Oxygen Level During Sleep
Description: Change from baseline in nadir oxygen level during sleep after a single dose of Venlafaxine will be evaluated using overnight polysomnography. A lower blood oxygen saturation during sleep is associated with a more severe obstructive sleep apnea.
Time Frame: Baseline and 7-day follow up
Measure: Median (Inter-Quartile Range); unit: Percent Oxygen Saturation
Arm/Group | Venlafaxine | Placebo
Number analyzed (Participants) | 20 | 20
Percent Oxygen Saturation | 82.0 [80.0 to 84.0] | 81.5 [75.8 to 84.2]

3. Secondary Outcome: Loop Gain
Description: Loop gain 1 is used to describe the stability of ventilatory control. The change from baseline in loop gain after a single dose of Venlafaxine will be estimated.
Time Frame: Baseline and 7-day follow up
Population: In one subject loop gain could not be quantified.
Measure: Mean (Standard Deviation); unit: Dimensionless
Arm/Group | Venlafaxine | Placebo
Number analyzed (Participants) | 19 | 19
Dimensionless | 0.58 (0.15) | 0.56 (0.14)

4. Secondary Outcome: Arousal Threshold
Description: Change from baseline in respiratory arousal threshold after single dose of Venlafaxine will be estimated.
Time Frame: Baseline and 7-day follow up
Population: In one subject arousal threshold could not be quantified.
Measure: Median (Inter-Quartile Range); unit: Percent V-eupnea
Arm/Group | Venlafaxine | Placebo
Number analyzed (Participants) | 19 | 19
Percent V-eupnea | 115.6 [108.2 to 130.8] | 118.6 [113.4 to 137.9]

5. Secondary Outcome: Sleep Efficiency
Description: Change from baseline in sleep efficiency after single dose of Venlafaxine will be estimated using overnight polysomnography.
Time Frame: Baseline and 7-day follow up
Measure: Mean (Standard Deviation); unit: Percent Time in Bed
Arm/Group | Venlafaxine | Placebo
Number analyzed (Participants) | 20 | 20
Percent Time in Bed | 63.1 (16.7) | 72.5 (15.5)

ADVERSE EVENTS:
Arm/Group | Venlafaxine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 2/20 | 1/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Venlafaxine (N=20) | Placebo (N=20)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) — Nausea without vomiting

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes